CLINICAL TRIAL: NCT07382414
Title: NUDGE-IHD: A Nationwide Pragmatic Randomized Trial of Electronic Nudges to Increase Patient Activation to Support Risk-factor Control in Ischemic Heart Disease
Brief Title: Electronic Letters to Improve Patient Activation in IHD: The NUDGE-IHD Trial
Acronym: NUDGE-IHD
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Tor Biering-Sørensen (Other)
Collaborators: Novartis (Industry)
Responsible Party: Sponsor-Investigator, Tor Biering-Sørensen, Professor, MD, MSc, MPH, PhD, Herlev and Gentofte Hospital
Organization: Herlev and Gentofte Hospital (Other)
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Health Services Research
Other Study IDs: F-24047871
Record Dates: First submitted 2025-12-09; First posted 2026-02-02 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: Coronary Artery Disease; Hypercholesterolemia; Lipoprotein(a); Secondary Prevention
MeSH Terms: conditions — Coronary Artery Disease; Hypercholesterolemia | interventions — Apolipoproteins A

STUDY DESIGN:
Intervention Model Description: Pragmatic, registry-based partial 2×2 factorial design.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- LDL letter only (Experimental): Participants randomized to the LDL-C letter but not the Lp(a) letter
  Interventions: Behavioral: LDL-C information letter
- Lp(a) letter only (Experimental): Participants randomized to the Lp(a) letter but not the LDL-C letter.
  Interventions: Behavioral: Lp(a) information letter
- No letter (No Intervention): Participants randomized to no LDL-C letter and to no Lp(a) letter
- LDL-C and Lp(a) letter (Experimental): Participants randomized to the LDL-C letter and the Lp(a) letter
  Interventions: Behavioral: LDL-C information letter; Behavioral: Lp(a) information letter

INTERVENTIONS:
Behavioral: LDL-C information letter — An electronically delivered informational letter communicating the participant's elevated LDL-C level and its relevance to ASCVD, with encouragement to consult their physician if relevant. Delivered via the Danish Digital Post system.
  Arms: LDL letter only; LDL-C and Lp(a) letter
Behavioral: Lp(a) information letter — An electronically delivered informational letter describing elevated Lp(a) as a genetically determined cardiovascular risk factor, with encouragement to discuss risk factor optimization with a physician if relevant.
  Arms: LDL-C and Lp(a) letter; Lp(a) letter only

SUMMARY:
The goal of this clinical trial is to learn whether simple electronic information letters can increase patient activation and improve risk-factor monitoring in adults in Denmark with ischemic heart disease (IHD) who have LDL cholesterol above the recommended treatment target. A subgroup of participants with elevated lipoprotein(a) [Lp(a)] will also be randomized to receive an additional information letter.

The main questions the study aims to answer are:

* Does sending an electronic letter about elevated LDL cholesterol increase the proportion of patients who have at least one LDL-cholesterol test within 6 months?
* Among patients with ischemic heart disease and elevated Lp(a), does receiving an information letter about Lp(a) increase patient activation, reflected by cardiometabolic risk-factor monitoring?

Because this is a randomized trial, researchers will compare people who receive the electronic letter(s) with people who do not receive any letter to determine whether the letters encourage patients to take action, such as obtaining laboratory tests or contacting their doctor.

Participants will:

* Receive an electronic letter through Denmark's national digital mailbox system (Digital Post) or receive no letter, depending on random assignment.
* Continue their usual health care, with no additional visits, treatments, or procedures required for the study.
* Have all study information collected from existing Danish nationwide health registries.

DETAILED DESCRIPTION:
This study is a nationwide, pragmatic, registry-based, partially factorial randomized trial conducted in Denmark. The trial evaluates whether simple electronic information letters ("nudges") can increase patient activation and support guideline-directed risk-factor monitoring among persons with ischemic heart disease (IHD) who have LDL cholesterol levels above guideline-recommended treatment targets in routine clinical care.

The primary study population consists of adults with documented ischemic heart disease and LDL cholesterol above the recommended target level. Eligible participants are identified using Danish nationwide health registries and randomized 1:1 to receive either an electronic information letter addressing elevated LDL cholesterol (the "LDL letter") or no letter. The LDL letter provides general, non-technical information about LDL cholesterol as a cardiovascular risk factor in ischemic heart disease and encourages recipients to consult their physician if relevant.

A secondary study population is defined as a subset of the primary population with elevated lipoprotein(a) [Lp(a)] levels identified from laboratory registry data. Participants in this subgroup are independently randomized 1:1 to receive or not receive an additional electronic information letter addressing elevated Lp(a) (the "Lp(a) letter"). The Lp(a) letter provides information on Lp(a) as a genetically determined and independent cardiovascular risk factor and emphasizes the importance of optimizing other modifiable risk factors. The two randomizations are conducted independently, resulting in a partially factorial design in which participants with elevated Lp(a) may receive no letter, the LDL letter only, the Lp(a) letter only, or both letters.

All intervention letters are delivered through Denmark's mandatory national digital mailbox system (Digital Post). The interventions are informational and non-invasive. The study does not involve any in-person visits, clinical procedures, or changes to usual medical care.

The primary outcome is disease-related patient activation, defined as the proportion of participants with at least one LDL cholesterol measurement recorded within 6 months after randomization. Secondary outcomes include general patient activation, assessed by the number of healthcare contacts in general practice or outpatient hospital settings, and cardiometabolic risk-factor monitoring, defined as the proportion of participants with at least one cardiometabolic blood test (lipid profile, hemoglobin A1c, or creatinine) within 6 months after randomization. Additional exploratory outcomes related to laboratory testing, healthcare utilization, medication use, and clinical events are assessed during longer-term follow-up.

All baseline characteristics, outcomes, and follow-up data are obtained from Danish nationwide health and administrative registries. Due to the registry-based and informational nature of the interventions, informed consent is not required. The primary analysis is conducted 6 months after randomization, with additional exploratory follow-up extending up to 5 years.

ELIGIBILITY:
Inclusion criteria

* Alive on identification date
* Diagnosis of IHD defined as either an A or B diagnosis code of I20-I25 in the Danish National Patient Register first registered > 6 months prior to identification date
* Latest available LDL-C is over 1.4 mmol/l measured up to 3 years prior to the identification date, defined using NPU codes NPU01568, NPU10171 or DNK35308 from the Danish National Laboratory Register
* Age >= 18 years and <= 85 on identification date

Exclusion criteria

* Nursing home residents
* Exemption from and thus not access to Digital Post

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100000 (Estimated)
Dates: Start 2026-04 (Estimated); Primary Completion 2026-10 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
the proportion of participants with at least one LDL-C measurement within 6 months following randomization | 6 months after randomization
  Whether the participant has at least one LDL-C laboratory measurement recorded in the Danish national laboratory registries within 6 months after randomization

SECONDARY OUTCOMES:
Number of healthcare contacts (general practice or outpatient hospital) within 6 months following randomization | 6 months after randomization
  Total number of healthcare contacts, defined as general practice contacts (in-person, telephone, or electronic) or outpatient hospital visits, recorded in national registries within 6 months after randomization.
At least one cardiometabolic blood test | Within 6 months after randomization
  Proportion of participants with at least one cardiometabolic blood test (lipid profile, hemoglobin A1c, or creatinine) recorded in Danish nationwide laboratory registries during follow-up.

CONTACTS AND LOCATIONS:
Locations (1):
- Center for Translational Cardiology and Pragmatic Randomized Trials, Department of Cardiology, Copenhagen University Hospital - Herlev and Gentofte, Hellerup, 2900, Hellerup, Region Sjælland, Denmark

IPD SHARING:
Plan to Share IPD: No
Data will be collected from Danish administrative health registries, which are subject to Danish legislation and can only be made available to a third party under certain conditions. Please contact the sponsor-investigator in case of any inquiries.